CLINICAL TRIAL: NCT03597191
Title: Effects of Spinal Stabilization Exercises on Dynamic Balance and Functional Performance in Adults With Subacute and Chronic Low Back Pain: A Randomized Clinical Trial
Brief Title: Effects of Spinal Stabilization Exercises on Dynamic Balance and Functional Performance in Adults With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Yousef Alshehre, Principal Investigator, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19982
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain; Chronic Low Back Pain; Subacute Low Back Pain
Keywords: Y-balance test; Functional Movement Screen; Spinal stabilization exercises; Dynamic balance; Postural control; Physical performance
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will be a randomized clinical trial (RCT) using a prospective two-way (2 × 4) mixed-design to examine the effectiveness of spinal stabilization exercises (SSEs) on dynamic balance, functional performance, pain intensity, and disability level in adults with sub-acute and chronic low back pain (LBP).
  The two independent variables are group, which is a between-subject factor, and time which is a within-subject factor. The independent variable of group has two levels: (1) the treatment group which will receive SSEs, and (2) the placebo group which will receive general range of motion and flexibility exercises.
  The independent variable of time has four levels: pre-intervention at baseline, and two weeks, four weeks, and eight weeks after intervention.
  The four dependent variables are (1) dynamic balance, (2) functional performance, (3) pain intensity, and (4) disability level.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The primary investigator (PI) of this study, the outcomes assessor, will be blinded to participants' group assignment and will perform the eligibility screening and standard physical therapy examination for all participants. In addition, the PI will perform the pre- and post-intervention measurements of dynamic balance using the Y- balance test, functional performance using Functional Movement Screen, pain scores using the Numeric Pain Rating Scale, and disability levels using the Modified Oswestry Low Back Pain Disability Questionnaire.
  Investigator #2, the care provider, will be blinded to the outcomes measurements and will be responsible for group allocation and administering the intervention, either a spinal stabilization exercises program or a general exercises program, to participants in both groups.
  Participants will be randomly assigned to one of the two study groups and will be blinded to the other group exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Stabilization Exercise Program (Experimental): Participants in the spinal stabilization exercise group will be instructed to perform four exercises in total, one exercise from each of the following four categories: (a) abdominal bracing, (b) quadruped, (c) prone plank, and (d) side plank exercises. Each exercise will be progressed and advanced in difficulty by increasing repetitions, hold times, and/or extremity movements.
  The progression of exercises will be based on the participants' performance at each supervised physical therapy session based on pre-established criteria by Hicks et al. (2005).
  Interventions: Other: Exercises
- General Exercises Program (Placebo Comparator): Participants in the general exercise group will perform a range of motion (ROM) and flexibility exercises of low back and lower extremities. Each participant will be instructed to perform four exercises in total, one exercise from each of the following four categories: (a) knee to chest, (b) lower trunk rotation, (c) prone press-ups, and (d) hamstring stretch exercises. These exercises will be progressed by increasing repetitions and pain-free ROM.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Participants in the treatment group will be instructed in the spinal stabilization exercises (SSEs), modeled after the spinal stabilization exercise program designed by Hicks et al. (2005). The SSE program targets muscle activation of spinal stabilizers specifically, the transversus abdominus and lumbar multifidus muscles. Each exercise will be progressed by increasing repetitions and hold time.

SUMMARY:
The investigators would like to know which one of two exercise programs will have a greater effect on balance, functional performance, daily function, and pain on individuals with low back pain (LBP) after 2, 4 and 8 weeks.

Specifically, the differences in dynamic balance, functional performance, pain intensity, and disability level will be compared between participants who receive spinal stabilization exercises program (SSE) and those who receive a general exercise program (GE) which includes range-of-motion (ROM) and flexibility exercises.

The research hypotheses are:

1. The SSE program will significantly improve dynamic balance and functional performance in adult participants with sub-acute and chronic LBP at two and four weeks as well as after an eight-week follow-up after initiating intervention.
2. The SSE program will significantly improve pain intensity and disability level in adult participants with sub-acute and chronic LBP at two and four weeks as well as after an eight-week follow-up after initiating intervention.
3. In adult participants with sub-acute and chronic LBP, the group receiving the SSE program will demonstrate significantly improved dynamic balance, functional performance, pain intensity and disability levels compared to the placebo group receiving the GE program at two and four weeks as well as after an eight-week follow-up after initiating intervention.

DETAILED DESCRIPTION:
Participants will be required to wear a pair of shorts, a loose T-shirt, and a pair of tennis shoes for this study. On the first visit, the investigators will do some tests to make sure that potential participant has good feeling and strength in his/her legs. Next, each participant will fill out a few forms asking about daily function and back pain. Then, the investigators will ask the participant to perform a balance test and seven functional tests. Two investigators will be there to give these tests.

During the balance test, each participant will stand on one leg and reach out for a distance with the other leg. During the functional tests, the participant will perform 7 different tasks, including a deep squat, hurdle step, in-line lunge, shoulder mobility, active straight leg raise, rotary stability and trunk stability push-up. The investigators will demonstrate these tests before the participant perform them.

After the balance and functional tests, each participant will be randomly assigned to one of the exercise programs. One of the investigators will instruct each participant to do the appropriate exercises depending on his/her ability and pain level.

After the first visit, participants will be asked to come back 1-2 times per week for 4 weeks so the investigators can update participants' exercise program and make sure that participants do each exercise in the correct form. Each follow-up visit will take about 30 minutes. In addition to the physical therapy visits, the investigators will ask participants to do the most updated exercises at home once a day and at least 5 times a week. The investigators will give each participant an exercise log to track the frequency of the home exercise sessions. At the end of the 4 weeks, participants will come to the last physical therapy session and will be asked to continue to do the updated exercises at home once a day and at least 5 times a week for another 4 weeks until the 8-week follow-up visit.

At the 2-week, 4-week and 8-week follow-up visit, the investigators will repeat the balance and the 7 functional tests.

Each testing session will last about 30 minutes. The testing sessions at 2 and 4 weeks will be done on the same visit of physical therapy for the participants' exercise sessions. During the 8-week follow-up visit, the investigators will ask the participants to fill out the forms about their daily function and back pain in addition to the balance and 7 functional tests. At the end of the 8 weeks, if the participants wish to have the other exercises, the investigators will instruct them with those exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the age of 18 to 65 years
2. Individuals who have low back pain (LBP) for 6 weeks or more
3. ability to understand, speak, and follow verbal instructions in English
4. the average pain level of at least 2 out of 10 in the past week

Exclusion Criteria:

1. serious spinal conditions such as fracture, infection, or tumor
2. signs of nerve root compression
3. a history of lower extremity or lumbar spine surgery
4. a history of hip, knee, or ankle pain in the previous two years
5. current pregnancy
6. systemic joint disease (e.g. rheumatologic or neurological disorders)
7. vestibular or other balance disorders
8. ongoing treatment for inner ear, sinus, or upper respiratory infection
9. concussion within the previous three months
10. a history of falls or fear of falling
11. a need for any form of walking aids (cane, walker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Change on dynamic balance | Change from baseline at two weeks, four weeks, and eight weeks post intervention.
  Dynamic balance measured by the Y-balance Test (YBT). Dynamic balance is quantified by measuring how far the reach indicator is placed relative to the stance platform while maintaining a unilateral stance. A farther reach distance is indicative of greater dynamic balance. To score each of the three directions, the reach distances (measured in cm) are averaged and normalized to the participant's leg length. As such, YBT scores are expressed as a percentage of leg length. Normalization is performed by dividing each reach distance by the participant's leg length and then multiplying by a hundred. Next, the composite score will be calculated by taking the average between right and left reach distances for all three directions and then summing the averages of the three reach directions. The score then will be divided by three times the average leg length and multiplied by 100.
Change on functional performance | Change from baseline at two weeks, four weeks, and eight weeks post intervention.
  Functional performance measured by Functional Movement Screen (FMS). Each participant will perform all 7 components of the FMS tests including deep squat, hurdle step, in-line lunge, shoulder mobility, active straight-leg-raise, trunk push-up, and trunk rotary stability tests. Participants will perform 3 trials for each of the 7 FMS tests, and the best score from the 3 trials will be recorded. In addition, each participant will perform 3 clearance screens. These 3 clearance screens evaluate pain and are graded as negative or positive. If a participant has no pain, the clearing test is considered negative. If there is an increase in pain, the clearing test is considered positive and the associated test will be scored zero. For movements that are scored on both limbs, the lower score will be used to compute the composite score. The total score of the 7 tests will be added together to get a composite score of the FMS.
Change on pain intensity level | Change from baseline at two weeks, four weeks, and eight weeks post intervention.
  pain intensity as perceived by the participant measured by the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point numerical scale (0-10), in which higher scores mean greater pain intensity. The possible scores on the NPRS range from zero representing no pain to 10 representing the worst imaginable pain. The NPRS will be administered verbally, and each participant will be asked to rate their pain intensity at present (i.e. current pain level).
Change on disability level | Change from baseline at two weeks, four weeks, and eight weeks post intervention.
  Modified Oswestry Low Back Pain Disability Questionnaire (OSW) to determine participants perceived disability level due to low back pain. The OSW is a self-reported ordinal scale measure that consists of 10 items assessing different aspects of pain and function related to the patient's LBP. Each item is scored on a six-point scale (0 to 5), with five representing the highest level of disability. The scores of the 10 items are then summed, with a maximum possible sum of 50 points. To obtain a percentage score, the sum is multiplied by two. Participants will be asked to use the OSW to rate their perceived level of disability at present.

SECONDARY OUTCOMES:
Fear-avoidance beliefs | at baseline and will be used for descriptive purposes only.
  To assess participants' beliefs regarding the effect of physical and work-related activities on their current LBP. The FABQ consists of 16 items and each item is scored on a seven-point Likert scale from zero (completely disagree) to six (completely agree), whereby higher scores indicate greater levels of fear-avoidance beliefs. This questionnaire comprises two independent subscales: the physical activity subscale which has five items (items1-5), and work subscale with eleven items (items 6-16). The participant should answer all items; however, for each subscale, not all items are included in the scoring. For scoring purposes, four items of the physical activity subscale are scored, with a possible score ranging from 0 to 24 points. Seven items of the work subscale are scored with a possible score ranging from 0 to 42 points. The five remaining FABQ items are not included in the score.
Patient Reported Outcomes Measurement Information System (PROMIS-29) | at baseline and will be used for descriptive purposes only.
  To characterize a range of participants' traits at baseline. The PROMIS-29 is a general health-related quality of life measure that assesses seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. In addition, pain intensity is measured with a single item on an 11-point numeric scale (NPRS) that ranges from 0 to 10. The PROMIS-29 scales will be scored using a T-score metric method available at the Assessment Center℠ website (http://assessmentcenter.net). Normative values have been reported for each domain of the PROMIS. As such, a score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean more of the specific scale's construct, which may indicate a desirable or an undesirable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yousef M Alshehre, MSc., Principal Investigator — Texas Woman's University; Khalid M Alkhathami, MPT, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's UniversityT. Boone Pickens Institute of Health Sciences-Dallas Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No